CLINICAL TRIAL: NCT06255665
Title: A Phase 1 Study of JNJ-79032421, a T-cell Redirecting Agent Targeting Mesothelin for Advanced Stage Solid Tumors
Brief Title: A Study of JNJ-79032421 Targeting Mesothelin for Advanced Stage Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109341; 79032421STM1001 (Other: Janssen Research & Development, LLC); 2023-504896-26-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Advanced Stage Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1 (Dose Escalation): JNJ-79032421 (Experimental): In Part 1 (Dose escalation), participants will receive JNJ-79032421. The dose will be escalated sequentially until the recommended phase 2 dose (RP2D) regimen(s) have been identified.
  Interventions: Drug: JNJ-79032421
- Part 2 (Dose Expansion): JNJ-79032421 (Experimental): In Part 2 (Dose expansion), participants will receive JNJ-79032421 at the RP2D regimen(s) determined in Part 1.
  Interventions: Drug: JNJ-79032421

INTERVENTIONS:
Drug: JNJ-79032421 — JNJ-79032421 will be administered.
  Arms: Part 1 (Dose Escalation): JNJ-79032421
Drug: JNJ-79032421 — JNJ-79032421 will be administered at RP2D regimen.
  Arms: Part 2 (Dose Expansion): JNJ-79032421

SUMMARY:
The purpose of this study is to determine recommended phase 2 dose(s) (RP2Ds) of JNJ-79032421 and to determine the safety and tolerability of JNJ-79032421 at the RP2D(s).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of one of the following unresectable/locally advanced or metastatic solid tumors: a) Ovarian cancer includes high grade serous epithelial ovary, fallopian tube, or primary peritoneal cancer. Participants must have progressed after at least 2 prior lines of systemic therapy and have either, i) platinum-refractory disease (ie, persistent disease following completion of platinum-based primary chemotherapy); or ii) platinum-resistant recurrent disease; b) Primary pleural or peritoneal mesothelioma. Sarcomatoid and well differentiated papillary histologies are not allowed. Participants must have progressed after at least 1 prior line of systemic therapy; c) Pancreatic ductal adenocarcinoma. Other histologies and mixed histologies are not allowed. Participants must have progressed after at least 1 prior line of systemic therapy.
* Measurable or evaluable disease: a) Part 1: Measurable or evaluable disease; b) Part 2: At least one measurable lesion per RECIST v1.1. Participants with mesothelioma must have disease measurable per mRECIST v1.1.
* Can have a prior or concurrent second malignancy (other than the disease under study) whose natural history or treatment is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1.
* Selected participants in the pharmacokinetic and pharmacodynamic (PK/PD) cohorts (Part 1) as well as selected participants in Part 2 must agree to undergo mandatory tumor biopsies.

Exclusion Criteria:

* History of known central nervous system (CNS) or leptomeningeal involvement.
* Left ventricular ejection fraction on screening echocardiogram below normal institutional limits.
* History of talc pleurodesis for pleural effusion within 3 months of starting study treatment.
* Concurrent empyema of the lung pleural space requiring antibiotics or chest tube or evidence of resultant fistula formation.
* History of hyperthermic intraperitoneal chemotherapy (HIPEC) within 6 months of starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicity (DLTs) | Up to first 21 days after first dose
  The DLTs are adverse events including certain high grade non-hematologic or hematologic toxicities, or toxicities meeting other specific criteria.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) by Severity | Up to 3 years
  An AE is any untoward medical occurrence in a clinical study participant administered an investigational or non-investigational product and it does not necessarily have a causal relationship with the investigational product. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome events (ICANS), which will be graded by American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.

SECONDARY OUTCOMES:
Part 1 and Part 2: Serum Concentration of JNJ-79032421 | Up to 3 years
  Serum concentration of JNJ-79032421 will be reported.
Part 1 and Part 2: Maximum Observed Analyte Concentration (Cmax) of JNJ-79032421 | Up to 3 years
  Cmax is defined as maximum observed analyte concentration of JNJ-79032421.
Part 1 and Part 2: Time to Reach Maximum Observed Analyte Concentration (Tmax) of JNJ-79032421 | Up to 3 years
  Tmax is defined as the time to reach maximum observed analyte concentration of JNJ-79032421.
Part 1 and Part 2: Area Under the Curve from Time t1 to Time t2 (AUC[t1-t2]) of JNJ-79032421 | Up to 3 years
  AUC(t1-t2) is defined as area under the analyte concentration for a specific time interval defined by t1 and t2 (AUC[t1-t2]) of JNJ-79032421.
Part 1 and Part 2: Number of Participants with Presence of Anti-JNJ-79032421 Antibodies | Up to 3 years
  The maximum titers of antibodies to JNJ-79032421 will be summarized for participants positive with antibodies to JNJ-79032421.
Part 1 and Part 2: Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as the percentage of participants with a best response of complete response or partial response according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1), and revised mRECIST for assessment of malignant pleural mesothelioma.
Part 1 and Part 2: Duration of Response (DOR) | Up to 3 years
  DOR is defined as the duration from the date of initial documentation of a response (PR or CR) to the date of first documented evidence of relapse or death according to RECIST v. 1.1, and revised mRECIST for malignant pleural mesothelioma.
Part 1 and Part 2: Cancer Antigen (CA) 125 Response Rate for Ovarian Cancer Only | Up to 3 years
  CA 125 response rate is defined as the proportion of participants with ovarian cancer who achieved a partial response or complete response according to the Gynecologic Cancer Intergroup (GCIG) response criteria for CA 125. A CA 125 response is defined as at least 50 percentage (%) reduction in CA 125 levels from a pretreatment sample which must be confirmed and maintained for at least 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- Spain (3):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency